CLINICAL TRIAL: NCT04533334
Title: Measurement of the Distance Between the Orifice of the Right Upper Lobe and Carinae and Labium Oris With Fiberoptic Bronchoscopy in Pediatric Population in Turkey
Brief Title: Measurement of the Distances of the Lower Airway in Pediatric Population
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kadir Melih YILMAZ, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 26082020
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Airway; Child; Bronchus
Keywords: anesthesia; fiberoptic bronchoscopy; lower airway anatomy; child; right upper lobe bronchus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric: FOB measurement of the distance between carina and right upper lobe bronchus and carina and labium oris in pediatric population
  Interventions: Procedure: FOB measurement

INTERVENTIONS:
Procedure: FOB measurement — A FOB will be inserted after anesthesia induction and the distances will be measured by direct observation via the bronchoscope.

SUMMARY:
Pediatric patients are exposed to increased risk during general anesthesia. A myriad of problems can be encountered in the pediatric population by misplaced endotracheal tubes. Especially, during one-lung ventilation (OLV) a right-sided or left-sided tube is inserted to facilitate the surgery. However, inadvertent tube use, caused by misinterpretation of the distances of the trachea and the main bronchi, may cause unintended hypoxemia, postoperative atelectasis and even mortality.

In this study, investigators will measure the distance between distal margin of right lung upper lobe orifice-carina and carina-lip with the help of fiberoptic bronchoscopy (FOB).

DETAILED DESCRIPTION:
In ASA-PS I-II-III children between 1-18 years of age who are orotracheally intubated for any reason, the fiber optic bronchoscope will be advanced in the tube and first the carina distance and then the carina to right upper bronchus distance will be measured.

Age, weight, height, body mass index (BMI), weight percentile, height percentile, comorbidities, ASA score, tube size, lip margin distance, right upper bronchus to carina distance and right upper lobe to carina distance/ Carina to-lip margin ratio will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing general anesthesia via an endotracheal tube
* ASA I-III

Exclusion Criteria:

* Patients that do not meet age criteria
* Uncontrolled asthma or hyper reactive airway
* hypoxemia, previous thoracic surgery
* ASA > III
* Unstable hemodynamics
* Patients with tracheal or oral malignancies
* Patients with face trauma
* Informed consent not given
* using a tube with a number too small for the fiberoptic bronchoscope to pass through

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients undergoing general anesthesia via an endotracheal tube will be eligible for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Upper/Lower Airway Ratio | 1 day
  Ratio of the distance between labium oris to carina and carina to right upper lobe orifice

SECONDARY OUTCOMES:
Correlation between patient characteristics and distances measured by FOB | 1 day
  Correlation between age, body mass index, gender, percentiles and the distance between labium oris to carina and carina to right upper lobe orifice

CONTACTS AND LOCATIONS:
Overall Officials: PINAR Kendigelen, MD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data available on reasonable request

REFERENCES:
- [Background] Rudraraju P, Eisen LA. Confirmation of endotracheal tube position: a narrative review. J Intensive Care Med. 2009 Sep-Oct;24(5):283-92. doi: 10.1177/0885066609340501. Epub 2009 Aug 3. PMID 19654121